CLINICAL TRIAL: NCT00880503
Title: Multidrug Resistance Molecular Target Analysis of Human Samples Collected in Clinical Trials Performed Outside of the Intramural National Cancer Institute
Brief Title: Collection of Tissue Samples for Study of Multidrug Resistance
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904067; 04-C-N067; NCT00898001 (obsolete NCT alias)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-02-08

CONDITIONS: Breast Carcinoma; Breast Cancer; Medullary Thyroid Carcinoma
Keywords: Multidrug Resistance Molecular Target Analysis
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Resistance to cancer chemotherapy develops in patients, rendering certain treatments ineffective. Despite much research, the prevailing cause of drug resistance is not known.

One mechanism for drug resistance involves a protein called P-glycoprotein, or Pgp, which reduces the effectiveness of cancer treatments by "pumping" anti-cancer drugs out of tumor cells where they are supposed to work against the disease.

Objectives:

To identify and evaluate more thoroughly the roles of Pgp and other substances in mediating drug resistance.

Eligibility:

Patients enrolled in clinical trials of cancer therapies at the Children's Hospital of Pittsburgh; Cancer Centers of Carolinas; Arizona Clinical Research Center; University of Copenhagen; and Herlev Hospital, Copenhagen who have consented to the use of blood, tissue, or tumor samples for laboratory studies.

Design:

Blood, tumor, and tissue samples are collected from participants and sent to the NCI for various laboratory analyses.

...

DETAILED DESCRIPTION:
Background:

Ultimately, patients who succumb to cancer do so because of drug resistance. Mechanisms of drug resistance have been explored in the laboratory and in clinical samples for some time, yet the prevailing cause of drug resistance, if indeed there is a single cause, is not known. One mechanism of drug resistance is multidrug efflux, mediated by P-glycoprotein. Other mechanisms have been proposed. Our laboratory has expertise in the analysis of drug transporter expression and activity in clinical samples.

Objectives:

To determine expression of P-glycoprotein and other multidrug transporters thought to mediate clinical drug resistance.

To evaluate inhibition of P-glycoprotein and other multidrug transporters through assessment of efflux activity in cells obtained from patients enrolled on clinical trials at other institutions.

To identify and evaluate mechanisms of drug resistance using molecular assays such as cDNA array, real-time PCR analysis, and immunohistochemistry.

Eligibility:

Patients enrolled on clinical trials outside the NCI, and giving informed consent to the use of blood, tissue, or tumor samples for evaluation of mechanisms of drug resistance or evaluation of inhibition of multi-drug efflux.

Future collaborations for similar studies will be added via the protocol amendment procedure; molecular studies other than ABC transporter assays will be added via the protocol amendment procedure.

Design:

Human tumor biopsies or blood samples will be collected from cancer patients enrolled on approved clinical trials, in accordance with the local protocol. These trials are being conducted at outside institutions, and the samples will be sent to the NCI for immunohistochemical analysis, cDNA array, PCR analysis, or for blood assays for detection of P-glycoprotein inhibition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patients entered on approved trials of cancer therapeutics at Children's Hospital of Pittsburgh, Herlev Hospital, and the University of Copenhagen outside of the intramural NCI are eligible for inclusion, provided that they have consented to tumor studies in the original consent forms.

EXCLUSION CRITERIA:

None anticipated at this time.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2003-12-19; Study Completion 2018-02-08

PRIMARY OUTCOMES:
Expression of MDR1/P-glycoprotein and related drug resistance proteins | Upon receipt and processing of specimen

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Childrens Hospital, Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Gottesman MM, Fojo T, Bates SE. Multidrug resistance in cancer: role of ATP-dependent transporters. Nat Rev Cancer. 2002 Jan;2(1):48-58. doi: 10.1038/nrc706. PMID 11902585
- [Background] Baer MR, George SL, Dodge RK, O'Loughlin KL, Minderman H, Caligiuri MA, Anastasi J, Powell BL, Kolitz JE, Schiffer CA, Bloomfield CD, Larson RA. Phase 3 study of the multidrug resistance modulator PSC-833 in previously untreated patients 60 years of age and older with acute myeloid leukemia: Cancer and Leukemia Group B Study 9720. Blood. 2002 Aug 15;100(4):1224-32. PMID 12149202
- [Background] Robey R, Bakke S, Stein W, Meadows B, Litman T, Patil S, Smith T, Fojo T, Bates S. Efflux of rhodamine from CD56+ cells as a surrogate marker for reversal of P-glycoprotein-mediated drug efflux by PSC 833. Blood. 1999 Jan 1;93(1):306-14. PMID 9864175